CLINICAL TRIAL: NCT05675566
Title: Investigation of Time-Dependent Change of Retention Force of Mandibular Implant Overdenture and Evaluation of Patient Satisfaction: A Clinical Follow-up Study
Brief Title: Time-dependent Change in the Retention Force of the Implant Overdenture
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ferit Bayram, Assist. Prof., Marmara University
Other Study IDs: MUDHF_PTT_01
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Edentulous Jaw
Keywords: Dental Prosthesis, Implant-Supported
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This descriptive longitudinal study aimed to investigate the retention force of implant-supported overdentures applied to edentulous individuals at Marmara University Faculty of Dentistry, examine the retention force and its time-dependent change, and evaluate patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 50-65 years old,
* Volunteer to participate in the study,
* Upper edentulous jaw with full denture, lower edentulous jaw with two-implant overdenture

Exclusion Criteria:

* Pregnant or lactating women
* Those who do not want to sign the consent form,
* Patients with a history of malignancy, radiotherapy, or chemotherapy
* Patients whose maxilla was rehabilitated with implant overdenture
* More than 2 implants for lower jaw implant overdenture

Ages: 50 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Our study will include individuals who have been rehabilitated with implant overdentures at Marmara University Faculty of Dentistry, Department of Prosthodontics.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change in retention force | 6 months
  The retention of a complete implant overdenture prosthesis is defined as the minimum retention force (N) required to separate the male part of the attachment from the female part. The retention strength will be measured 3 times with a force gauge that allows the application of the retention force perpendicular to the occlusal plane of the prosthesis and parallel to the long axis of the implant, and the values will be averaged with a digital dynamometer. As the measurement value increases, it is concluded that the retention of the prosthesis increases. The measurements will be recorded on the 'Patient Measurement Card' at each control session.
  The retention of the implanted complete denture will be measured at the time of delivery of the implant overdenture to the patient and at the control sessions 1 week, 1 month, 3 months, and 6 months after the patient start to use the denture.

SECONDARY OUTCOMES:
Change in patient satisfaction | 6 months
  Patients' overall satisfaction, comfort, speech ability, prosthesis stability, retention, aesthetics, and ease of cleaning will be assessed using VAS measurements. The rating words will be 'very satisfied' and 'not at all satisfied,' and patients will be asked to draw a vertical line on a 10 cm horizontal line at the point that best represents their perception. The VAS total score is between 0-10. As the score increases, it is concluded that the patient's satisfaction increases. Patients will be asked to fill out the VAS questionnaire form during the 1st month (TI) after using the prosthesis and at 3 months and 6 months of control sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Akoglu B, Ucankale M, Ozkan Y, Kulak-Ozkan Y. Five-year treatment outcomes with three brands of implants supporting mandibular overdentures. Int J Oral Maxillofac Implants. 2011 Jan-Feb;26(1):188-94. PMID 21365055
- [Background] Cousson PY, Bessadet M, Nicolas E, Veyrune JL, Lesourd B, Lassauzay C. Nutritional status, dietary intake and oral quality of life in elderly complete denture wearers. Gerodontology. 2012 Jun;29(2):e685-92. doi: 10.1111/j.1741-2358.2011.00545.x. Epub 2011 Oct 17. PMID 22004061
- [Background] Evtimovska E, Masri R, Driscoll CF, Romberg E. The change in retentive values of locator attachments and hader clips over time. J Prosthodont. 2009 Aug;18(6):479-83. doi: 10.1111/j.1532-849X.2009.00474.x. Epub 2009 Jun 3. PMID 19500236
- [Background] Fromentin O, Lassauzay C, Abi Nader S, Feine J, de Albuquerque Junior RF. Testing the retention of attachments for implant overdentures - validation of an original force measurement system. J Oral Rehabil. 2010 Jan;37(1):54-62. doi: 10.1111/j.1365-2842.2009.02020.x. Epub 2009 Nov 11. PMID 19912482
- [Background] Sultana N, Bartlett DW, Suleiman M. Retention of implant-supported overdentures at different implant angulations: comparing Locator and ball attachments. Clin Oral Implants Res. 2017 Nov;28(11):1406-1410. doi: 10.1111/clr.13003. Epub 2017 Feb 13. PMID 28191678
- [Background] Ucankale M, Akoglu B, Ozkan Y, Ozkan YK. The effect of different attachment systems with implant-retained overdentures on maximum bite force and EMG. Gerodontology. 2012 Mar;29(1):24-9. doi: 10.1111/j.1741-2358.2010.00389.x. Epub 2010 Jun 30. PMID 20604812
- [Background] Uludag B, Polat S, Sahin V, Comut AA. Effects of implant angulations and attachment configurations on the retentive forces of locator attachment-retained overdentures. Int J Oral Maxillofac Implants. 2014 Sep-Oct;29(5):1053-7. doi: 10.11607/jomi.3401. PMID 25216129